CLINICAL TRIAL: NCT00086307
Title: Combining a Dopamine Agonist and Selective Serotonin Reuptake Inhibitor for Treatment of Depression: A Double-Blind, Randomized Study
Brief Title: Lexapro and Pramipexole and to Treat Major Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Carlos Zarate, M.D., Chief of Experimental Therapeutics and Pathophysiology Branch of NIMH, DIRP, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 040227; 04-M-0227
Record Dates: First submitted 2004-06-29; First posted 2004-06-30 (Estimated); Results first posted 2012-07-12 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Major Depression
Keywords: Pramipexole; Escitalopran; Antidepressant; Dopaminergic Receptor Agonist; Depression; Major Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Pramipexole; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pramipexole (Active Comparator): Patients receive pramipexole and placebo. The dosage of pramipexole is 0.125 milligrams (mg) three times per day in the first week, 0.250 mg three times per day in the second week, 0.5 mg three times per day in the third week, and 0.75 mg three times per day in the fourth week and thereafter.
  Interventions: Drug: Pramipexole
- Escitalopram (Active Comparator): Patients receive escitalopram and placebo. The dosage of escitalopram is 10 milligrams (mg) per day.
  Interventions: Drug: Escitalopram
- Escitalopram and Pramipexole (Experimental): Patients receive escitalopram and pramipexole. The dosage of escitalopram is 10 milligrams (mg) per day. The dosage of pramipexole is 0.125 mg three times per day in the first week, 0.250 mg three times per day in the second week, 0.5 mg three times per day in the third week, and 0.75 mg three times per day in the fourth week and thereafter.
  Interventions: Drug: Pramipexole; Drug: Escitalopram

INTERVENTIONS:
Drug: Pramipexole — Pramipexole will be titrated so patients receive the following medication three times per day during the weeks noted: .125 milligrams (mg) in week 1, .250 mg in week 2, .5 mg in week 3, and .75 mg in weeks 4 to 6.
  Arms: Escitalopram and Pramipexole; Pramipexole
Drug: Escitalopram — Escitalopram will be started at 10 mg/day and patients will continue on this throughout the study.
  Arms: Escitalopram; Escitalopram and Pramipexole

SUMMARY:
This study compares the effectiveness of the combination of antidepressants: Lexapro and Pramipexole, with the effectiveness of each antidepressant alone.

Purpose: Patients between 18 and 65 years of age with Major Depressive Disorder without psychotic features may be eligible for this 9-week study. Candidates must currently be in a major depressive episode of at least 4 weeks' duration, have failed to respond to treatment with an SSRI (Prozac, Zoloft, Paxil, Luvox, Celexa), and not have failed to respond to more than four antidepressants for the current episode. Candidates are screened with a physical examination, psychiatric evaluation, blood tests, review of vital signs, height and weight measurements, electrocardiogram (ECG), urine test for illegal drugs, and pregnancy test for women.

Participants are tapered off antidepressants or other medications prohibited during the study and remain drug-free for 1 week before starting treatment. They are then randomly assigned to take pramipexole and escitalopram, pramipexole alone, or escitalopram alone for 6 weeks. During the study, participants come to the clinic eight times for health assessments and symptoms assessments, which include a check of vital signs and rating scales for depression and anxiety, adverse events, and sexual functioning. Blood and urine samples are collected periodically to monitor health, detect pregnancy in women, and detect illicit drug use.

At the end of the 6-week treatment period, participants have a physical examination, ECG, blood test, and check of vital signs. Short-term anti-depressant treatment is offered, and plans are made for long-term treatment.

Atendemos pacientes de habla hispana.

...

DETAILED DESCRIPTION:
Despite the availability of a wide range of antidepressant drugs, 30% to 40% of patients with major depression fail to respond to first-line antidepressant (e.g., selective serotonin reuptake inhibitors [SSRIs]) treatment, despite adequate dosage, duration, and compliance. Furthermore, these medications may take weeks to months to achieve their full effects, and in the meantime, patients continue to suffer from their symptoms and continue to be at risk of self-harm as well as harm to their personal and professional lives. Thus, there is a clear need to develop novel and improved therapeutics for treatment-resistant major depression that are more effective and have a rapid onset of action. Preclinical and clinical studies suggest that antidepressants with a combined mechanism of action (e.g., combination of a selective serotonin-reuptake inhibitor (SSRI) and a norepinephrine reuptake inhibitor) may be more effective than either agent alone in achieving remission (Nelson et al 2004). Thus, it stands to reason that other combinations of antidepressants with other mechanisms of action when combined may have a synergistic effect that is superior to an antidepressant with a single mechanism of action. Preclinical and clinical studies suggest that the dopaminergic system may play a major role in the pathophysiology of depression. Preclinical studies suggest synergistic antidepressant effects with the combination of a SSRI and a selective D3 receptor agonist in animal models of depression. Similarly, preliminary clinical studies suggest synergism with combination treatment that affects the serotonin and dopamine systems. Together, these data suggests that treatments which affect the serotonin and dopamine systems will be more effective than agents which use a single mechanism. We propose to compare the combination of a selective dopaminergic agonist and a SSRI in patients with treatment-resistant major depression. To our knowledge, this will be the only controlled double-blind study to date that will examine the efficacy of a serotonin and dopamine combination given from the start of treatment.

Patients, ages 18 years or older, with a diagnosis of major depression (without psychotic features), will be randomized to the combination of a selective dopaminergic receptor agonist and a SSRI or either drug alone for a period of 6 weeks. Acute efficacy will be determined by demonstrating a greater remission rate using specified criteria. Approximately 115 patients with acute major depression will be enrolled in the study.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Male or female subjects, 18 to 65 years of age.
2. Female subjects of childbearing potential must be using a medically accepted means of contraception.
3. Each subject must have a level of understanding sufficient to agree to all required tests and examinations and sign an informed consent document.
4. Subjects must fulfill DSM-IV criteria for Major Depression (296.33) without psychotic features, based on clinical assessment and confirmed by a structured diagnostic interview, SCID-P.
5. Subjects must have an initial score of greater than or equal to 20 on the MADRS at Visit 1 and Visit 2.
6. Subjects must not have a greater than a 25% decrease in the MADRS total scores during washout (between Visits 1 and 2).
7. Current or past history of lack of response to at least one adequate antidepressant trial (SSRI) operationally defined using the Antidepressant Treatment History Form (ATHF) (Sackeim 2001b). If this criteria has not been met, a four-week prospective trial of a standard antidepressant (at the patients' and clinicians' discretion) may be given. Subjects are excluded if greater than four failed antidepressant trials for the current major depressive (adequate dose and duration as defined by the ATHF).
8. Current major depressive episode of at least 4 weeks duration.

   EXCLUSION CRITERIA:
9. Presence of psychotic features or a diagnosis of Schizophrenia or any other psychotic disorder or bipolar disorder as defined in the DSM-IV.
10. Subjects with a history of DSM-IV drug or alcohol dependency or abuse (except for nicotine or caffeine) within the preceding 3 months.
11. Previously failed to respond to an adequate trial (dose and duration) of escitalopram.
12. Female subjects who are either pregnant or nursing.
13. Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
14. Subjects with uncorrected hypothyroidism or hyperthyroidism.
15. Subjects with one or more seizures without a clear and resolved etiology.
16. Previous treatment with pramipexole.
17. Treatment with a reversible MAOI within 2 weeks prior to Visit 2.
18. Treatment with fluoxetine within 5 weeks prior to Visit 2.
19. Treatment with any other concomitant medication not allowed (Appendix A) 7 days prior to study Visit 2.
20. Treatment with clozapine or ECT within 3 months prior to study Visit 2.
21. Judged clinically to be an acute suicidal risk.
22. Psychotherapy will not be permitted during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Zarate, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Agnoli A, Ruggieri S, Casacchia M. Restatement and prospectives of ergot alkaloids in clinical neurology and psychiatry. Pharmacology. 1978;16 Suppl 1:174-88. doi: 10.1159/000136818. No abstract available. PMID 347463
- [Background] Anderson IM. SSRIS versus tricyclic antidepressants in depressed inpatients: a meta-analysis of efficacy and tolerability. Depress Anxiety. 1998;7 Suppl 1:11-7. PMID 9597346
- [Background] Agren H, Mefford IN, Rudorfer MV, Linnoila M, Potter WZ. Interacting neurotransmitter systems. A non-experimental approach to the 5HIAA-HVA correlation in human CSF. J Psychiatr Res. 1986;20(3):175-93. doi: 10.1016/0022-3956(86)90002-6. PMID 2430098

RESULTS

PARTICIPANT FLOW:
Groups:
- Pramipexole: Patients receive pramipexole and placebo.
- Escitalopram: Patients receive escitalopram and placebo.
- Escitalopram and Pramipexole: Patients receive escitalopram and pramipexole.
Period: Overall Study
Arm/Group | Pramipexole | Escitalopram | Escitalopram and Pramipexole
Started | 13 | 13 | 13
Completed | 11 | 12 | 5
Not Completed | 2 | 1 | 8
Not completed — Lack of Efficacy | 1 | 1 | 2
Not completed — Shortness of breath and muscle spasms | 1 | 0 | 0
Not completed — Nausea and headaches | 0 | 0 | 1
Not completed — Constipation and sleepiness | 0 | 0 | 1
Not completed — Suicidal ideation | 0 | 0 | 1
Not completed — Fatigue and difficulty falling asleep | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pramipexole | Escitalopram | Escitalopram and Pramipexole | Total
Number analyzed (Participants) | 13 | 13 | 13 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 13 | 39
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 44.8 (10.1) | 45.6 (13.6) | 45.3 (12.7) | 45.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 11 | 27
  Male | 6 | 4 | 2 | 12
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 13 | 39

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Rating Scale (MADRS)
Description: The Montgomery Asberg Depression Rating Scale (MADRS) is a 10 item scale for assessing the severity of depression. Items are rated on a scale of 0 to 6, so the maximum score is 60 and the minimum is 0, where 60 is the most severe depression. Scores of 18 or greater are generally considered to indicate a moderate level of depression.
Time Frame: Weekly
Population: All patients with at least one post-baseline measurement were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Pramipexole | Escitalopram | Escitalopram and Pramipexole
Number analyzed (Participants) | 13 | 13 | 13
Score on a scale | 22.629 (1.508) | 26.102 (1.507) | 29.455 (1.732)
Statistical Analysis 1: Comparison: Pramipexole vs Escitalopram vs Escitalopram and Pramipexole; A linear mixed model with restricted maximum likelihood estimation and a first order autoregressive covariance structure was used to examine depressive symptoms over time. Fixed factors for drug, time, and a time by drug interaction were included in the model along with the intercept. No random factors were included because the subject factor did not contribute significantly to the model. Baseline symptoms were used as a covariate; Test type: Superiority or Other; p = .018, Mixed Models Analysis — This is the omnibus effect of drug; Mean Difference (Net) = 6.826, 95% CI 2-sided [1.111 to 12.541], Standard Error of Mean 2.296
Statistical Analysis 2: Comparison: Pramipexole vs Escitalopram and Pramipexole; Post-hoc simple effects tests with Bonferroni correction were used to compare the pramipexole group to the pramipexole and escitalopram combination group; Test type: Superiority or Other; p = .014, Post hoc simple effects test — The significance level was adjusted using a Bonferroni correction; Mean Difference (Net) = 6.826, 95% CI 2-sided [1.111 to 12.541], Standard Error of Mean 2.296 — The pramipexole group had a lower MADRS score than the pramipexole and escitalopram group
Statistical Analysis 3: Comparison: Escitalopram vs Escitalopram and Pramipexole; Post-hoc simple effects tests with Bonferroni correction were used to compare the escitalopram group to the pramipexole and escitalopram combination group; Test type: Superiority or Other; p = .454, Post hoc simple effects test — The significance level was adjusted using a Bonferroni correction; Mean Difference (Net) = 3.353, 95% CI 2-sided [-2.360 to 9.066], Standard Error of Mean 2.296 — The escitalopram group had a lower MADRS score than the pramipexole and escitalopram group
Statistical Analysis 4: Comparison: Pramipexole vs Escitalopram; Post-hoc simple effects tests with Bonferroni correction were used to compare the pramipexole group to the escitalopram group; Test type: Superiority or Other; p = .349, Post hoc simple effects test — The significance level was adjusted using a Bonferroni correction; Mean Difference (Net) = 3.473, 95% CI 2-sided [-1.942 to 8.888], Standard Error of Mean 2.162 — The pramipexole group had a lower MADRS score than the escitalopram group

ADVERSE EVENTS:
Arm/Group | Pramipexole | Escitalopram | Escitalopram and Pramipexole
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 8/13 | 12/13 | 11/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pramipexole (N=13) | Escitalopram (N=13) | Escitalopram and Pramipexole (N=13)
Headache (General disorders) | 3 (3) | 3 (3) | 4 (4)
Dizziness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Eye Irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Earache (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Dry Mouth (General disorders) | 0 (0) | 1 (1) | 1 (1)
Nasal Congestion (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sore Throat (General disorders) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Ailment (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
Nausea (General disorders) | 3 (3) | 1 (1) | 5 (5)
Vomiting (General disorders) | 1 (1) | 0 (0) | 1 (1)
Constipation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (General disorders) | 2 (2) | 1 (1) | 1 (1)
Stool Discoloration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Appetite Increase (General disorders) | 0 (0) | 3 (3) | 2 (2)
Appetite Decrease (General disorders) | 1 (1) | 1 (1) | 4 (4)
Increased Thirst (General disorders) | 1 (1) | 2 (2) | 1 (1)
Painful Urination (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Increased Frequency of Urination (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Menstrual Irregularity (Reproductive system and breast disorders) | 1/7 (1) | 0/9 (0) | 1/11 (1)
Premenstrual Tension (Reproductive system and breast disorders) | 0/7 (0) | 1/9 (1) | 0/11 (0)
Increased Libido (General disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased Libido (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sexual Dysfunction (General disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle/Bone/Joint Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 3 (3)
Tic Movements (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatological Irritation (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Hair Problems (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (3) | 0 (0)
Increased Motor Activity (General disorders) | 0 (0) | 0 (0) | 2 (2)
Decreased Motor Activity (General disorders) | 1 (1) | 0 (0) | 0 (0)
Difficulty Falling Asleep (General disorders) | 0 (0) | 1 (1) | 5 (5)
Early Morning Awakening (General disorders) | 0 (0) | 2 (2) | 4 (4)
Interrupted Sleep (General disorders) | 1 (1) | 2 (2) | 3 (3)
Drowsiness (General disorders) | 0 (0) | 4 (4) | 0 (0)
Slurred Speech (General disorders) | 0 (0) | 0 (0) | 1 (1)
Concentration Difficulty (General disorders) | 0 (0) | 1 (1) | 2 (2)
Memory Problems (General disorders) | 1 (1) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (3) | 4 (4)
Irritability (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Suicidal Ideas (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Breast pain or swelling (Skin and subcutaneous tissue disorders) | 1/7 (1) | 0/9 (0) | 0/11 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Accidental injury (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No